CLINICAL TRIAL: NCT07140224
Title: Korfball-Based Training and Motor Skill Development in Young Athletes: A Randomized Trial
Brief Title: Korfball-Based Training and Motor Skill Development
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Gaziantep (Other)
Responsible Party: Principal Investigator, Burak Karaca, Mr., University of Gaziantep
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 2025/04
Record Dates: First submitted 2025-08-18; First posted 2025-08-24 (Actual); Last update posted 2025-08-29 (Actual); Status verified 2025-08

CONDITIONS: Motor Skills Development; Physical Fitness; Physical Education and Training/Methods
Keywords: korfball; explosive power; mixed-gender training; youth sports; physical education

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The investigators conducting the outcome measurements were blinded to group assignments and study hypotheses to reduce bias.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): Control group continued with their usual school-based physical education classes without any additional training (8 week).
- Korfball Training Group (Experimental): The korfball training group participated in an eight-week korfball-based movement training program, three times a week, each session lasting 90 minutes. Training consistently occurred from 16:00 to 18:00 in an outdoor korfball court under coach supervision. Each session started with 10 minutes of warming up and 5 minutes of stretching exercises. The main session included 65 minutes of korfball-based movement training, followed by a 10-minute cool-down period.
  Interventions: Other: Korfball-Based Movement Training

INTERVENTIONS:
Other: Korfball-Based Movement Training — The weekly training content was structured as follows:
  * Week 1: Chest pass, overhead pass, right-left hand pass, moving pass, cool-down (15 repetitions).
  * Week 2: One-handed pass, penalty shot, defensive follow-up run, lay-up shot, cool-down (20 repetitions).
  * Week 3: One-handed pass, diagonal passing, penalty shot, lay-up shot, short and long-distance shooting (25 repetitions).
  * Week 4: Lay-up shot, V-cut shot, stationary short-distance shot, defensive follow-up run,penalty shot, cool-down (20 repetitions).
  * Week 5: V-cut shot, stationary short-distance shot, front-of-the-basket shot, behind-the-basket short-distance shot (15 repetitions).
  * Week 6: V-cut shot, lay-up shot, stationary shot, defensive follow-up run, penalty shot (20 repetitions).
  * Week 7: One-handed pass, penalty shot, lay-up shot (right-left), shooting, V-cut shot (10 repetitions).
  * Week 8: One-handed pass penalty shot, lay-up shot (right-left), stationary shot, V-cut shot (10 repetitions).
  Arms: Korfball Training Group

SUMMARY:
The goal of this randomized trial is to find out if an 8-week korfball-based training program can improve lower-body strength and jumping ability in children aged 10-12 years. Korfball is a mixed-gender sport that promotes teamwork and equal participation.

The study will test two main questions:

Does korfball training increase explosive leg power measured by the Margaria-Kalamen Stair Climb Test? Does korfball training improve performance in the Standing Long Jump Test?

Children are randomly assigned to one of two groups:

Korfball Training Group: Participants take part in supervised korfball-based exercise sessions 3 times per week for 8 weeks, in addition to their normal school activities.

Control Group: Participants continue with standard school physical education classes only.

All participants complete both the Margaria-Kalamen Stair Climb Test and the Standing Long Jump Test before and after the 8-week period.

This study will show whether korfball training is an effective and inclusive way to improve explosive leg power and motor skills in school-aged children.

DETAILED DESCRIPTION:
Korfball is a mixed-gender team sport that emphasizes cooperation, spatial awareness, and technical ball skills. Its unique format prohibits gender-based physical contact and requires players to coordinate offensive and defensive movements in a cooperative way. These characteristics make korfball not only a socially inclusive activity but also a potential tool for motor development in children. However, there is limited experimental evidence examining the physical benefits of korfball training in youth populations.

This randomized controlled trial was designed to investigate whether an 8-week korfball-based training program can improve explosive lower-body performance in children aged 10-12 years. A total of 30 participants were randomly assigned to either a korfball training group or a control group. The training group completed three 90-minute sessions per week for eight weeks, in addition to their regular school physical education classes. The control group continued with their standard school-based activities only.

The intervention program included structured korfball drills such as passing, shooting, lay-up techniques, and defensive footwork. Sessions were organized progressively from basic skills to more complex game-like movements. All training sessions were supervised by a certified physical education teacher to ensure safety and protocol fidelity.

Two validated physical performance tests were used to assess outcomes:

Margaria-Kalamen Stair Climb Test (MK): to evaluate anaerobic power by measuring the time taken to ascend stairs with predetermined step intervals.

Standing Long Jump Test (SLJ): to assess horizontal explosive power of the lower limbs.

Tests were conducted before and after the 8-week intervention under standardized conditions. Trained evaluators blinded to group assignments recorded all measurements. The primary outcome was change in Margaria-Kalamen test performance, while the secondary outcome was change in Standing Long Jump distance.

The study hypothesis was that participants in the korfball training group would demonstrate significantly greater improvements in both MK and SLJ performance compared to the control group, regardless of gender. By testing this hypothesis, the trial aims to provide evidence for korfball as a safe, inclusive, and effective training method for improving lower-limb explosive strength in school-aged children.

If positive, the findings could inform physical education curricula and youth sports programming, supporting the use of korfball-based activities as a practical approach to enhance motor development while promoting gender equality in sport participation.

ELIGIBILITY:
Inclusion Criteria:

* Healthy children aged 10-12 years
* Regular participation in school-based physical activity or physical education classes
* Ability to attend training sessions and testing procedures for the full 8-week - period
* Written informed consent obtained from parents/guardians

Exclusion Criteria:

* Presence of chronic or acute illnesses (e.g., cardiovascular, respiratory, or metabolic diseases)
* Orthopedic or musculoskeletal injuries/disorders that may limit safe participation
* Neurological disorders affecting motor performance
* Lack of regular participation in physical activities prior to study enrollment
* Failure to obtain parental/guardian consent

Ages: 10 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 30 (Actual)
Dates: Start 2025-05-01 (Actual); Primary Completion 2025-06-26 (Actual); Study Completion 2025-06-27 (Actual)

PRIMARY OUTCOMES:
Margaria-Kalamen Stair Climb Test (Explosive Power) | Baseline (pre-test) and after 8 weeks of training (post-test)
  Change in anaerobic power output (watts) measured using the Margaria-Kalamen stair climb test. Participants sprinted up a staircase stepping on the 3rd, 6th, and 9th steps. Anaerobic power was calculated using the standard formula P = (m × g × h) / t, where m is body mass (kg), g is gravitational acceleration (9.81 m/s²), h is the vertical height between the 3rd and 9th steps (1.2 m), and t is the time taken to ascend (s).
Standing Long Jump Test (Horizontal Explosive Power) | Baseline (pre-test) and after 8 weeks of training (post-test)
  Change in horizontal jump distance (cm) measured using the Standing Long Jump test. Participants jumped forward from a standing start with both feet together, and the best of three trials was recorded.

CONTACTS AND LOCATIONS:
Locations (1):
- Gaziantep University, Gaziantep, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data (IPD) underlying the results (e.g., test scores from Margaria-Kalamen and Standing Long Jump) will be available upon reasonable request from the corresponding author. De-identified datasets may be shared for academic research purposes only, following approval by the principal investigator and in compliance with data protection regulations.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: De-identified individual participant data (IPD) and supporting documents will be available beginning 6 months after publication of the study results and will remain accessible for 5 years thereafter.
Access Criteria: De-identified individual participant data (IPD), including test results from the Margaria-Kalamen Stair Climb Test and the Standing Long Jump Test, as well as supporting documents (Study Protocol, Statistical Analysis Plan, Informed Consent Form), will be available to qualified academic researchers. Data will be shared solely for non-commercial, academic research purposes upon reasonable request to the corresponding author. Requests will be reviewed by the principal investigator to ensure compliance with ethical standards and data protection regulations. Access will be granted through secure data transfer after approval.